CLINICAL TRIAL: NCT06421350
Title: Efficacy of Closed-Loop Spinal Cord Stimulation for Complex Regional Pain Syndrome
Brief Title: Closed Loop Spinal Cord Stimulation for Complex Regional Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, David Hiller, MD, Principal Investigator, Scripps Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-8347
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Acute and Subacute Phases of CRPS (Experimental): Participants diagnosed with acute and subacute phases of CRPS will be assigned to this group.
  Interventions: Device: Spinal Cord Stimulation Device
- Chronic Phase of CRPS (Experimental): Participants diagnosed with chronic CRPS will be assigned to this group.
  Interventions: Device: Spinal Cord Stimulation Device

INTERVENTIONS:
Device: Spinal Cord Stimulation Device — The closed-loop spinal cord stimulation mechanism uses dynamic adjusting stimulation parameters based on real-time physiologic response and is uniquely positioned to mitigate the aberrant inflammatory and neurosensory processing and autonomic dysfunction driving CRPS and its progression between phases.

SUMMARY:
The primary purpose of this study is to determine the differences in response to treatment of complex regional pain syndrome with a closed-loop spinal cord stimulator if applied in the early phases (acute or subacute) versus the chronic phase.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, all patients given written informed consent will be organized into group 1 (acute or subacute) and group 2 (chronic). They will undergo a trial period with a temporary spinal cord stimulator for 7 days. After the trial period, if the provider determines the device improved the patient's pain and function, the permanent device will be implanted. The patient will fill out an outcomes packet at baseline, end of trial period, 3 months and 6 months. There will also be a blood draw to evaluate prolactin levels, which are associated with stress and pain, at baseline, end of trial period, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* neuromodulation naive patients with unilateral CRPS type 1 or type 2 (defined by Budapest Criteria)
* pre-procedure psychological clearance

Exclusion Criteria:

* younger than 18 years
* prior neuromodulation including spinal cord stimulation
* prior dorsal root ganglion stimulation
* prior peripheral nervous system stimulation
* anatomical obstacles to dorsal column lead placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Complex Regional Pain Syndrome Severity Scores | Baseline, 7 day trial period, 3 months, 6 months
  (CRPS SS) This will be determined at baseline by the provider based on his diagnosis of the patient's condition, being acute and subacute or chronic. This is based on the presence or absence of 16 clinically-assessed signs and symptoms, and complements the diagnostic criteria for CRPS. A higher score indicates greater severity of the condition. This will be followed up at the 7 day trial period, 3 months and 6 months post procedure by evaluation.
Change in Target Activation Amplitude Levels by the Spinal Cord Stimulation Device | 7 day trial period, 3 months, and 6 months.
  Spinal cord stimulation device parameters will be collected to determine if a lower voltage is required to treat acute phase of complex regional pain syndrome as compared to later phases. This will be conducted at follow up visits and analyzed by the medical device representative. The data will be pulled and analyzed to determine the activation point for each patient. This will be captured at the 7 day trial period, 3 months, and 6 months.

SECONDARY OUTCOMES:
Change in Prolactin Levels | Baseline, 7 day trial period, and 3 months
  We plan to include a physiological marker of pain response by assessing serum prolactin levels, which are linked to dopamine levels in the brain. We will use prolactin as a convenient marker of abnormal dopamine levels due to chronic pain and the response to spinal cord stimulation treatment as an objective quantifiable metric of success with treatment. We will collect this via blood draw at our lab at baseline, at the 7 day trial period, and 3 months.
Visual Analogue Pain Scale | Baseline, 7 day trial period, 3 months, and 6 months
  (VAS) This will be used to determine the pain intensity the patient is experiencing. It will be on a scale from 0-10, 0 being no pain and 10 being the worst pain.
Quality of Life Questionnaire | Baseline, 7 day trial period, 3 months, and 6 months
  (EQ-5D-5L) Used to capture quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A lower score would indicate a severe score and the patient has a low quality of life. The patient also rates how good or bad their health is on a scale of 0-100, 100 being the best health and 0 being the worst health they could imagine.
Patient Reported Outcomes Measurement Information System-29 v 2.1 | Baseline, 7 day trial period, 3 months, and 6 months
  (PROMIS-29v2.1) Used to assess pain intensity using a single 0-10 numeric rating item and seven health domains: physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance.
General Anxiety Disorder-7 | Baseline, 7 day trial period, 3 months and 6 months.
  (GAD-7) Used for the screening and severity measuring of generalized anxiety disorder. It consists of seven items the patients rate based on their experiences over the past two weeks. Each item is scored from 0 (none) to 3 (every day). The cumulative score, ranging from 0-21, indicates the severity of GAD symptoms, with higher scores corresponding to greater anxiety levels.
Patient Health Questionnaire-9 | Baseline, 7 day trial period, 3 months, 6 months
  (PHQ-9) Used for screening and measuring the severity of depression. A higher score would indicate the patient has a worse outcome.
Short-Form McGill Pain Questionnaire-2 | Baseline, 7 day trial period, 3 months, 6 months
  (SF-MPQ-2) Used to rate the intensity of each type of pain and related symptoms. A higher score means the patient has a worse outcome. They rate their pain and symptoms on a scale of 0-10, with a 0 being no pain and 10 being the worst pain.
Pain Catastrophizing Scale | Baseline, 7 day trial period, 3 months, 6 months
  (PCS) Used to assess catastrophic thinking related to pain among adults with or without chronic pain. A higher score would mean the patient has a worse outcome.
Patient Global Impression of Change | 7 day trial period, 3 months and 6 months
  (PGIC) Used to measure the patient's belief about the effectiveness of the treatment. A higher score would reflect the patient believes the treatment is not effective and they have been doing much worse.
Amount of Pain Medication Consumed by Patient | Baseline, 7 day trial period, 3 months and 6 months
  Used to track amount of pain medication taken by the patient on a daily basis or what they are taking and when they are taking it.

CONTACTS AND LOCATIONS:
Overall Officials: David B Hiller, MD, Principal Investigator — Physician
Locations (1):
- Scripps Clinic Torrey Pines, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No